CLINICAL TRIAL: NCT05046054
Title: The Effect of Transcutaneous Electrical Nerve Stimulation on Pain During Propofol Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-03-036-001
Record Dates: First submitted 2021-09-05; First posted 2021-09-16 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Transcutaneous Electrical Nerve Stimulation; Pain; Propofol Adverse Reaction
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: TENS YW-5000 (YoungWon Medical Co, Korea)
Who Masked: Investigator
Masking Description: Two electrodes were attached to the radial side of dominant forearm. In the placebo group the TENS device had no current output although the power "on" indicator light remained active.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous electrical nerve stimulation group (Active Comparator): Transcutaneous electrical nerve stimulation was givent via two electrodes on the venous cannulation site 20 min before propofol injection
  Interventions: Device: transcutaneous electrical nerve stimulation
- control group (Placebo Comparator): No transcutaneous electrical nerve stimulation was not given via two electrodes on the venous cannulation site 20 min before propofol injection
  Interventions: Device: Placebo transcutaneous electrical nerve stimulation

INTERVENTIONS:
Device: transcutaneous electrical nerve stimulation — transcutaneous electrical nerve stimulation group received transcutaneous electrical nerve stimulation via two electrodes on the venous cannulation site 20 min before propofol injection
  Arms: transcutaneous electrical nerve stimulation group
Device: Placebo transcutaneous electrical nerve stimulation — Placebo transcutaneous electrical nerve stimulation group received no transcutaneous electrical nerve stimulation via two electrodes on the venous cannulation site 20 min before propofol injection
  Arms: control group

SUMMARY:
Propofol, an intravenous sedative agent, frequently produces pain during injection. This study was designed to investigate whether transcutaneous electrical nerve stimulation could reduce pain during propofol injection.

in minimizing propofol injection pain.

DETAILED DESCRIPTION:
Twenty min after transcutaneous electrical nerve stimulation, the electrodes were removed and propofol 0.5 mg/kg was administered at the rate of 0.5 ml/sec using syringe pump. Propofol injection pain was evaluated by a study blinded anesthesiologist using a four point scale: 0=no (negative response to questioning), 1=mild pain (pain reported only in response to questioning without any behavioral sings), 2=moderate pain (pain reported in response to questioning and accompanied by a behavioral signs or pain reported spontaneously without questioning, 3=severe pain (strong vocal response or response accompanied by facial grimacing, arm withdrawal or tears).

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* American Society of Anesthesiologists physical status classification > 3
* Patient with a history of allergy to drugs
* Patient who takes opioid, sedative, anticonvulsant
* Patient with a history of neurologic disease and psychological disorders
* patient with skin problem
* Patient with pacemaker or electric medical device
* pregnancy

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
pain during propofol injection | 15 seconds
  Propofol injection pain was evaluated by a study blinded anesthesiologist using a four point scale

CONTACTS AND LOCATIONS:
Overall Officials: Younghoon Jeon, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National university hospital, Daegu, South Korea